CLINICAL TRIAL: NCT06498128
Title: QUVIVIQ® Pregnancy Registry
Brief Title: Registry to Collect Information on Pregnancy, Neonatal, and Infant Outcomes in Pregnant Women Exposed to QUVIVIQ®
Status: Recruiting | Type: Observational
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: ID-078A403; 1000000033 (Other: Catalogue of RWD studies)
Record Dates: First submitted 2024-06-17; First posted 2024-07-12 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Insomnia
Keywords: Pregnancy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — daridorexant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 21 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- QUIVIQ (Cohort A): Women with insomnia exposed to QUVIVIQ during pregnancy or within 5 half-lives prior to conception.
  Interventions: Drug: Daridorexant
- Non-orexin receptor antagonist medications for insomnia (Cohort B1): Women exposed to other, non-orexin receptor antagonist medications for insomnia during pregnancy or within 5 half-lives of the respective insomnia medication prior to conception.
  Interventions: Drug: Non-orexin receptor antagonist medications for insomnia
- No insomnia medications (Cohort B2): Women who had no exposure to any insomnia medication during pregnancy and within 5 half-lives of any insomnia medication taken prior to conception.
  Interventions: Other: No insomnia medication

INTERVENTIONS:
Drug: Daridorexant — Dosing and treatment duration of QUVIVIQ as part of this observational study is at the discretion of the healthcare provider in accordance with local clinical practice and local labeling.
  Other Names: QUVIVIQ
  Groups: QUIVIQ (Cohort A)
Drug: Non-orexin receptor antagonist medications for insomnia — Dosing and treatment duration of non-orexin receptor antagonist medications for insomnia as part of this observational study is at the discretion of the healthcare provider in accordance with local clinical practice and local labeling.
  Groups: Non-orexin receptor antagonist medications for insomnia (Cohort B1)
Other: No insomnia medication — No insomnia medication was administered.
  Groups: No insomnia medications (Cohort B2)

SUMMARY:
This study will investigate pregnancy, neonatal, and infant outcomes in women exposed to QUVIVIQ during pregnancy compared to women unexposed to QUVIVIQ during pregnancy.

ELIGIBILITY:
A) Eligibility criteria for prospective pregnancies:

Inclusion Criteria:

1. Diagnosis of insomnia disorder prior to pregnancy.
2. Pregnancy is ongoing and outcome of pregnancy (i.e., pregnancy loss or live birth) is not known.
3. One of the following:

   1. Exposure to QUVIVIQ at any time during the current pregnancy or within 5 half-lives prior to conception.
   2. Exposure to other, non-orexin receptor antagonist medications for insomnia during pregnancy or within 5 half-lives of the respective insomnia medication prior to conception.
   3. No exposure to any insomnia medication during pregnancy and within 5 half-lives of any insomnia medication taken prior to conception.

Exclusion Criteria:

* Exposure to any orexin receptor antagonist other than QUVIVIQ - including BELSOMRA® (suvorexant), DAYVIGO® (lemborexant), any orexin receptor antagonist newly approved during the study period, or any orexin receptor antagonist in pre-market clinical studies - during the current pregnancy or within 5 half-lives of the respective medication prior to conception.

B) Eligibility criteria for retrospective pregnancies:

Inclusion criteria:

1. Diagnosis of insomnia disorder prior to pregnancy.
2. Pregnancy has ended.
3. Exposure to QUVIVIQ during pregnancy or within 5 half-lives prior to conception.

Exclusion criteria:

* Exposure to any orexin receptor antagonist other than QUVIVIQ - including suvorexant, lemborexant, any orexin receptor antagonist newly approved during the study period, or any orexin receptor antagonist in pre-market clinical studies - during pregnancy or within 5 half-lives of the respective medication prior to conception.

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Women with insomnia disorder, monitored in a standard-of-care setting, and pregnant at time of enrollment (prospective pregnancies) will be assigned to a specific cohort according to the insomnia medication received. Women with insomnia disorder for whom the outcome of pregnancy is known prior to enrollment (retrospective pregnancies) will be analyzed in a separate case series.
Sampling Method: Non-Probability Sample
Enrollment: 785 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2033-03 (Estimated); Study Completion 2033-03 (Estimated)

PRIMARY OUTCOMES:
Major congenital malformations classified according to MACDP | Start of pregnancy up to 1 year of infant age
  Congenital malformations will be classified according to the Metropolitan Atlanta Congenital Defects Program (MACDP) classification system. All potential major congenital malformations identified by the participant's or the infant's healthcare providers will be evaluated by a qualified, independent committee of at least 3 teratologists using all available medical records. Classification will be based upon the teratologists' adjudication, who will be blinded to participant exposure status.

SECONDARY OUTCOMES:
Pregnancy complications - number of participants with pre-eclampsia | 20 weeks gestation until delivery/birth/labor
  The presence of hypertension on 2 occasions at least 4 hours apart after 20 weeks gestation (in a woman with previously normal blood pressure) and proteinuria; or, in the absence of proteinuria, a new onset of hypertension accompanied by one of the following conditions: thrombocytopenia, renal insufficiency, impaired liver function, pulmonary edema, or cerebral or visual symptoms.
Pregnancy complications - number of participants with pregnancy-induced hypertension | 20 weeks gestation until delivery/birth/labor
  High blood pressure associated with pregnancy, as diagnosed by the treating healthcare provider, i.e., elevated (systolic between 120-129 mmHg and diastolic less than 80 mmHg); Stage 1 hypertension (systolic between 130-139 mmHg or diastolic between 80-89 mmHg); or Stage 2 hypertension (systolic at least 140 mmHg or diastolic at least 90 mmHg).
Pregnancy complications - number of participants with pre-term labor | Start of pregnancy up to 37 weeks gestation
  Regular contractions of the uterus resulting in changes in the cervix that start before 37 weeks of pregnancy.
Pregnancy complications - number of participants with gestational diabetes | Start of pregnancy until delivery/birth/labor
  Characterized by the development of carbohydrate intolerance with first onset or first recognition during pregnancy.
Pregnancy outcomes - number of participants with pregnancy outcome of elective or therapeutic pregnancy termination | Start of pregnancy until delivery/birth/labor
  Any induced or voluntary fetal loss during pregnancy.
Pregnancy outcomes - number of participants with pregnancy outcome of spontaneous abortion | Start of pregnancy up to 20 weeks gestation
  Loss of a fetus due to natural causes at less than 20 weeks of gestation.
Pregnancy outcomes - number of participants with pregnancy outcome of fetal death or stillbirth | 20 weeks gestation up to birth
  Death of a fetus at or after 20 weeks of gestation.
Pregnancy outcomes - number of participants with pregnancy outcome of live birth | 37 weeks gestation up to 40 weeks gestation
  Birth of a surviving neonate.
Pregnancy outcomes - number of participants with pregnancy outcome of pre-term birth | Less than 34 weeks gestation up to 37 weeks gestation
  Live birth prior to 37 weeks gestation: early preterm (< 34 weeks), late preterm (34-36 weeks), and early term (37-38 weeks).
Infant outcomes - number of infants with outcome of minor congenital malformations classified according to MACDP | Start of pregnancy up to 1 year of infant age
  Congenital malformations will be classified according to the Metropolitan Atlanta Congenital Defects Program (MACDP) classification system. All potential minor congenital malformations will be evaluated by at least 3, qualified, independent teratologists using all available medical records. Classification will be based upon the teratologists' adjudication, who will be blinded to participant exposure status.
Infant outcomes - infants categorized according to size for gestational age | At birth of infant
  All live births will be classified using the World Health Organization definition of birth weight, i.e., small (below the 10th percentile), appropriate (between the 10th and 90th percentile), or large (above the 90th percentile) for gestational age.
Infant outcomes - number of infants with outcome of low birth weight | At birth of infant
  Birth weight of less than 2500 g; subclassified into very low birth weight (< 1500 g) and moderately low birth weight (1500 g to 2499 g).
Infant outcomes - number of infants with outcome of infant death | Birth of infant up to 1 year of infant age
  Death of a live-born infant within the first year of life; subclassified as neonatal deaths (≤ 28 days of life) and infant deaths (29 to 365 days of life).
Infant outcomes - number of infants with outcome of hospitalization for serious illness | Birth of infant up to 1 year of infant age
  In-patient admissions for treatment of potentially life threatening illnesses among live-born infants within the first year of life.
Infant outcomes - postnatal growth and development - weight-for-length | Birth of infant up to 1 year of infant age
  World Health Organization Growth Charts (suitable for use in the US and EEA from birth to 24 months) will be applied for this study, where infant growth measurements will be used to estimate gender-specific weight-for-length percentiles (weight in kilograms, length in centimeters).
Infant outcomes - postnatal growth and development - head circumference-for-age | Birth of infant up to 1 year of infant age
  World Health Organization Growth Charts (suitable for use in the US and EEA from birth to 24 months) will be applied for this study, where infant growth measurements will be used to estimate gender-specific head circumference-for-age percentiles (head circumference in centimeters, age in months and years).
Infant outcomes - postnatal growth and development - length-for-age | Birth of infant up to 1 year of infant age
  World Health Organization Growth Charts (suitable for use in the US and EEA from birth to 24 months) will be applied for this study, where infant growth measurements will be used to estimate gender-specific length-for-age percentiles (length in centimeters, age in months and years).
Infant outcomes - postnatal growth and development - weight-for-age | Birth of infant up to 1 year of infant age
  World Health Organization Growth Charts (suitable for use in the US and EEA from birth to 24 months) will be applied for this study, where infant growth measurements will be used to estimate gender-specific weight-for-age percentiles (weight in kilograms, age in months and years).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials Study Director, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (7):
- IQVIA US Office, Durham, North Carolina, United States
- Jodha Tishon, Toronto, Ontario, Canada
- Hôpital Gui de Chauliac, Montpellier, France
- Charité - Universitätsmedizin Berlin, Berlin, Germany
- Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Rome, Italy
- Hospital Txagorritxu, Vitoria-Gasteiz, Spain
- University College London Hospitals, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No